CLINICAL TRIAL: NCT06651528
Title: An Innovative, Trauma-informed Approach for Reducing Overdose Risk Among Women Re-entering the Community From Prison
Brief Title: Trauma-informed Intervention to Reduce Substance Use and to Support Community Transition
Acronym: TRUST
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Michele Staton (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Michele Staton, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94956; R33DA061365 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-21 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: Overdose; Criminal legal system; Trust-based relational intervention (TBRI)
MeSH Terms: conditions — Substance-Related Disorders; Drug Overdose | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment As Usual (TAU) (Active Comparator): Traditional in-prison SUD treatment
  Interventions: Other: Treatment as Usual (TAU)
- TRUST only (Experimental): Treatment as usual and the adapted version of TBRI for adult women (TRUST Intervention)
  Interventions: Behavioral: TAU + TRUST
- TRUST + Re-entry Recovery Support (Experimental): Treatment as usual, the adapted intervention (TRUST), and on-going re-entry recovery support with the Safe Support Person (SSP).
  Interventions: Behavioral: TAU + TRUST + Re-entry Recovery Support

INTERVENTIONS:
Behavioral: TAU + TRUST — The adapted TBRI WRA (Prison Only Component) titled TRUST will consist of an individual introductory module (1 hour) and a series of group modules (a minimum of 4 sessions, approximately 1-2 hours in length, delivered over the course of 3 months, with the final number and frequency to be determined in R61) focused on the core components of TBRI. The original TBRI approach includes a focus on group skills training; similarly, it is anticipated that R61 phase adaptations will meet the need for tailored skills training reflected by anticipated differences in the target population of women - including how their early attachment and trauma histories influence their current self-image and behavior (which likely has a tremendous impact on their relational attachments as adults). Group sessions will provide opportunities to build skills for regulating emotions and building healthy connections.
  Arms: TRUST only
Behavioral: TAU + TRUST + Re-entry Recovery Support — This condition includes the proposed adapted TRUST intervention as well as on-going re-entry recovery support with the Safe Support Person (SSP). The SSP will be identified by the study participant as someone who will provide prosocial support during re-entry (e.g., support towards abstinence, establishing healthy recovery support relationships, rebuilding relationships with family and children) and in most cases will involve a close family member (mother, grandmother) or friend at the woman's identified home placement. This individual will be identified by the study participant as someone who is not involved in active substance use nor has a current legal system status (e.g., on probation).
  Arms: TRUST + Re-entry Recovery Support
Other: Treatment as Usual (TAU) — Women in the TAU condition will not receive TRUST intervention services, but will receive traditional in-prison SUD treatment over 6 months as usual in the four targeted prison sites. The programs are separate units with the prisons and emphasize participation by all program members in the overall goal of addressing substance use and criminal thinking. Although trauma and violence are addressed as part of the holistic group process approach in these programs, these topics are not addressed from an on-going systematic or relational perspective and are not specifically addressed as part of re-entry planning.
  Arms: Treatment As Usual (TAU)

SUMMARY:
The overall aim of this study is to reduce overdose risk for criminal legal system (CLS) involved women during community re-entry through the adaptation and testing of an innovative, trauma-informed, relational intervention approach (Trust-Based Relational Intervention or TBRI).

DETAILED DESCRIPTION:
R61 Phase (Intervention adaptation): The TBRI intervention will be strategically adapted for CLS-involved women during the R61 to achieve 2 specific aims: 1) Adapt TBRI by focusing on adapting two intervention components - prison group sessions and re-entry recovery support - using focus groups with key stakeholders (N=30) including administrators, practitioners, and women with "lived experience," and target alignment with the unique treatment needs of the women and establish intervention approach feasibility; and 2) Pilot test the adapted intervention components in one group of women (n=8) at the KCIW facility. Final adaptations will be made to the TRUST manual for the R33 implementation.

R33 Phase (Intervention testing): The R33 will test the effectiveness of the adapted TBRI-WRA to reduce overdose risk in the community following prison release, while also collecting data on key constructs hypothesized to influence successful intervention implementation. The primary aim of the R33 is to examine effectiveness of the adapted TBRI Women's Re-entry Approach (TBRI-WRA) in reducing overdose risk among women (N=264) in four sites following release from prison-based SUD treatment. Study conditions include (1) Treatment as Usual (TAU, standard in-prison SUD treatment, n=88), (2) In-prison TBRI (TAU + TBRI prison-based sessions only; n=88), and (3) TBRI + Re-entry Recovery Support (TAU + prison-based TBRI sessions + Re-entry Recovery Support; n=88). The R33 will also examine implementation factors associated with study preparation, launch, sustainability, and scalability.

ELIGIBILITY:
Inclusion Criteria:

* participating in corrections-based SUD treatment
* have an anticipated parole eligibility date within 4 months
* self-identified history of violent victimization
* are willing to work with at least one person living in the community who will be supportive of your recovery when you get out
* interested in participating in the study

Exclusion Criteria:

* not participating in corrections-based SUD treatment
* anticipated parole eligibility date greater than 4 months
* no self-identified history of violent victimization
* not willing to work with at least one person living in the community who will be supportive of your recovery when you get out
* not interested in participating in the study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Change in overdose risk | Baseline and at 3 and 6 months post-release from prison
  Change in number of days of any substance from baseline to post-release using self-report data

SECONDARY OUTCOMES:
Change in trauma-related symptoms | Baseline and at 3 and 6 months post-release from prison
  Change in number of trauma-related symptoms associated with violence

CONTACTS AND LOCATIONS:
Overall Officials: Michele Staton, MSW, PhD, Principal Investigator — University of Kentucky; Kevin Knight, PhD, Principal Investigator — Texas Christian University
Locations (4):
- United States (4):
  - Franklin County Regional Jail, Frankfort, Kentucky
  - Kentucky Correctional Institution for Women, Pewee Valley, Kentucky
  - Chillicothe Correctional Center, Chillicothe, Missouri
  - Women's Eastern Reception, Diagnostic and Correctional Center, Vandalia, Missouri

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.